CLINICAL TRIAL: NCT05786924
Title: A Phase 1/2, Open-label Study of Oral S241656 (BDTX-4933) as Monotherapy and in Combination With Other Anti-Cancer Therapies in Patients With KRAS, BRAF and Other Selected RAS/MAPK Mutation-Positive Malignancies
Brief Title: Phase 1/2 Trial of S241656 in Selected RAS/MAPK Mutation- Positive Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BDTX-4933-101; 2025-523474-16-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-06; First posted 2023-03-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer; Histiocytic Neoplasm; Histiocytosis; BRAF Gene Mutation; BRAF V600E; BRAF V600 Mutation; BRAF Mutation-Related Tumors; BRAF; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Lung Cancer; Recurrent Lung Cancer; Recurrent Lung Non-Small Cell Carcinoma; NSCLC; Solid Tumor; Solid Carcinoma; KRAS G12D; KRAS G12V; KRAS Mutation-Related Tumors; NRAS Gene Mutation; Thyroid Cancer; Thyroid Carcinoma; Colorectal Cancer; Colorectal Carcinoma; Recurrent Histiocytic and Dendritic Cell Neoplasm; Brain Metastases; Recurrent NSCLC; KRAS G13C; Acquired Resistance to KRAS G12C Inhibitor; KRAS G12A; KRAS G12F; KRAS G12R; KRAS G13D
Keywords: BRAF Class I; BRAF Class II; BRAF Class III; KRAS; Intolerant histiocytic neoplasm; BDTX-4933; Phase 1; dose escalation; dose expansion; MAPK; mitogen-activated protein kinase; RAS; RAF; Upstream oncogenic alterations; RAF inhibitor; intracranial disease; CRAF; NRAS; RAF fusions
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Histiocytosis; Lung Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms; Brain Neoplasms | interventions — IFL protocol; Cetuximab; Panitumumab; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Part 1A: Dose Escalation NSCLC (Experimental): S241656 will be administered as a monotherapy at escalating dose levels until the biologically effective dose (BED) range is determined.
  Interventions: Drug: S241656
- Part 1B: Dose Escalation GI Tumors (Experimental): S241656 will be administered as a monotherapy at escalating dose levels until the BED range is determined.
  Interventions: Drug: S241656
- Part 1C: Dose Escalation PDAC (Experimental): S241656 will be administered in combination with gemcitabine/nab-paclitaxel at escalating dose levels until the BED range is determined.
  Interventions: Drug: S241656; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Part 1D: Dose Escalation CRC (Experimental): S241656 will be administered in combination with FOLFOX6/FOLFOX7 or FOLFIRI, and panitumumab or cetuximab at escalating dose levels until the BED range is determined.
  Interventions: Drug: S241656; Drug: FOLFOX6/FOLFOX7; Drug: FOLFIRI; Drug: Cetuximab; Drug: Panitumumab
- Part 1E: Dose Escalation Other Solid Tumors (Experimental): S241656 will be administered as a monotherapy at escalating dose levels until the BED range is determined.
  Interventions: Drug: S241656
- Part 2A: Dose Optimization NSCLC (Experimental): S241656 will be administered to further characterize the optimal dose.
  Interventions: Drug: S241656
- Part 2A1: Dose Expansion NSCLC with KRAS non-G12C mutations (Experimental): S241656 will be administered as a monotherapy in the BED range.
  Interventions: Drug: S241656
- Part 2A2: Dose Expansion NSCLC with BRAF mutations (Experimental): S241656 will be administered as a monotherapy in the BED range.
  Interventions: Drug: S241656
- Part 2A3: Dose Expansion NSCLC with KRAS non-G12C or BRAF mutations/alterations (Experimental): S241656 will be administered as a monotherapy in the BED range. Participants must also have active CNS metastatic disease
  Interventions: Drug: S241656
- Part 2A4: Dose Expansion NSCLC with a KRAS G12C mutation (Experimental): S241656 will be administered as a monotherapy in the BED range. Participants must have received and progressed upon G12C targeted therapy
  Interventions: Drug: S241656
- Part 2B1: Dose Expansion PDAC (Experimental): S241656 will be administered as a monotherapy in the BED range.
  Interventions: Drug: S241656
- Part 2B2: Dose Expansion CRC (Experimental): S241656 will be administered as a monotherapy in the BED range.
  Interventions: Drug: S241656
- Part 2B3: Dose Expansion BTC (Experimental): S241656 will be administered as a monotherapy in the BED range.
  Interventions: Drug: S241656
- Part 2C1: Dose Expansion PDAC (Experimental): S241656 will be administered in combination with anti-cancer therapies in the BED range. The combination therapies to be used will be determined in the future.
  Interventions: Drug: S241656
- Part 2D1: Dose Expansion CRC (Experimental): S241656 will be administered in combination with anti-cancer therapies in the BED range. The combination therapies to be used will be determined in the future.
  Interventions: Drug: S241656
- Part 2F: Exploratory Food Effect (Experimental): S241656 will be administered as a monotherapy.
  Interventions: Drug: S241656

INTERVENTIONS:
Drug: S241656 — RAF inhibitor targeting all classes of oncogenic BRAF alterations (Classes I, II, and III) and constitutively active CRAF, KRAS or NRAS mutations
  Other Names: BDTX-4933
Drug: FOLFOX6/FOLFOX7 — Used as a combination therapy and administered intravenously
  Arms: Part 1D: Dose Escalation CRC
Drug: FOLFIRI — Used as a combination therapy and administered intravenously
  Arms: Part 1D: Dose Escalation CRC
Drug: Cetuximab — Used as a combination therapy and administered intravenously
  Arms: Part 1D: Dose Escalation CRC
Drug: Panitumumab — Used as a combination therapy and administered intravenously
  Arms: Part 1D: Dose Escalation CRC
Drug: Gemcitabine — Used as a combination therapy and administered intravenously
  Arms: Part 1C: Dose Escalation PDAC
Drug: Nab-paclitaxel — Used as a combination therapy and administered intravenously
  Arms: Part 1C: Dose Escalation PDAC

SUMMARY:
BDTX-4933-101 is a first-in-human, open-label, Phase 1/2 dose escalation, dose optimization and expansion study designed to evaluate the safety and tolerability of S241656 as monotherapy and in combination with other anti-cancer therapies in participants with selected advanced malignancies. The study population for the Dose Escalation part of the study comprises adults with recurrent advanced/metastatic non-small cell lung cancer (NSCLC), Gastrointestinal (GI) cancers, and other solid tumors harboring KRAS, HRAS, NRAS, BRAF, and/or CRAF (Rapidly Accelerated Fibrosarcoma (RAF1)) mutations or alterations. A dose optimization part in adults with NSCLC may follow the dose escalation phase if the sponsor, in consultation with the safety review committee, decides it is necessary to further characterize the optimal dose. However, the study may also proceed directly to the expansion phase. The study population for the Dose Expansion part of the study comprises adults with advanced/metastatic NSCLC with KRAS and/or BRAF mutations, and with Pancreatic Ductal AdenoCarcinoma (PDAC), ColoRectal Cancer (CRC), and Biliary Tract Cancer (BTC) with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations and alterations. All patients will self-administer S241656 orally in 28-day cycles until disease progression, toxicity, withdrawal of consent, or termination of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Life expectancy of ≥ 12 weeks in the opinion of the investigator.
* Histologically or cytologically confirmed recurrent locally advanced (unresectable) or metastatic solid tumors with documented RAS or RAF mutations or alterations.
* Adequate bone marrow and organ function.
* Recovered from toxicity to prior anti-cancer therapy.

Part 1 Dose Escalation cohort ONLY:

* Part 1A: Advanced/metastatic NSCLC with KRAS non-G12C, HRAS, NRAS, BRAF or CRAF (RAF1) mutations or alterations
* Part 1B: Advanced/metastatic GI tumors (e.g., PDAC, CRC, and BTC) with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations or alterations
* Part 1C: Advanced/metastatic PDAC with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations or alterations
* Part 1D: Colorectal adenocarcinoma with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations or alterations
* Part 1E: Other advanced/metastatic non-GI, non-NSCLC solid tumors with KRAS, HRAS, NRAS, BRAF, CRAF (RAF1) mutations or alterations

Part 2 Dose Optimization and Expansion cohorts ONLY:

* Part 2A: Advanced/metastatic NSCLC with KRAS non-G12C mutations and/or BRAF mutations
* Part 2A1: Advanced/metastatic NSCLC with KRAS non-G12C mutations
* Part 2A2: Advanced/metastatic NSCLC with BRAF mutations
* Part 2A3: Advanced/metastatic NSCLC with KRAS non-G12C or BRAF mutations or alterations and active CNS metastatic disease
* Part 2A4: Advanced/metastatic NSCLC with a KRAS G12C mutation
* Part 2B1: Advanced/metastatic PDAC with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations or alterations
* Part 2B2: Advanced/metastatic CRC with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations or alterations
* Part 2B3: Advanced/metastatic BTC (adenocarcinoma) with KRAS, HRAS, NRAS, BRAF, and/or CRAF (RAF1) mutations or alterations

Key Exclusion Criteria:

* Cancer that has a known MEK1/2 mutation.
* Known allergy/hypersensitivity to excipients of S241656 or to any of the registered IMPs administered in combination.
* Any contra-indication, to use of any of the combination chemotherapy or anti-EGFR therapy partners administered as part of this trial.
* Major surgery within 4 weeks of study entry or planned during study.
* Ongoing anticancer therapy.
* Ongoing radiation therapy.
* Uncontrolled or active clinically relevant bacterial, fungal, or specific viral infection requiring systemic therapy.
* Clinically significant cardiovascular disease.
* Symptomatic spinal cord compression.
* Evidence of active malignancy (other than study-specific malignancies) requiring systemic therapy within the next 2 years.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO.
* Females who are pregnant or breastfeeding.
* Actively receiving systemic treatment or direct medical intervention on another therapeutic clinical study.
* Prior use of experimental agents that target the KRAS/BRAF/MEK/ERK pathway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of dose-limiting toxicities (DLTs) | The first 28-day cycle (Cycle 1)
  A DLT is defined as any event meeting the DLT criteria occurring within the first 28-day cycle
Dose Escalation: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, approximately 5 years
Dose Optimization/Expansion: Objective response (OR) | Through study completion, approximately 5 years

SECONDARY OUTCOMES:
Dose Escalation/Expansion: Incidence and severity of treatment-emergent adverse events (TEAEs) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Maximum plasma concentration (Cmax) of S241656 and its metabolite S243796 | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Time of maximum plasma concentration (Tmax) of S241656 and its metabolite S243796 | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Area under the plasma drug concentration-time curve (AUC) of S241656 and its metabolite S243796 | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Half-life (t1/2) of S241656 and its metabolite S243796 | Through study completion, approximately 5 years
Dose Escalation: Objective response (OR) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Disease Control (DC) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Clinical Benefit (CB) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Duration of response (DOR) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Time to response (TTR) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Progression-free Survival (PFS) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Overall survival (OS) | Through study completion, approximately 5 years
Dose Optimization/Expansion: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Number of Dose Interruptions | Through study completion, approximately 5 years
Dose Escalation/Optimization/Expansion: Number of Dose Reductions | Through study completion, approximately 5 years
Dose Escalation: Number of Dose Discontinuations | Through study completion, approximately 5 years
Dose Optimization/Expansion: Changes in allelic fraction of DNA sequence variants detected in ctDNA from baseline to on-treatment time points | Through study completion, approximately 5 years

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Banner Health- MD Anderson Cancer Center, Gilbert, Arizona
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - Georgetown University Lombardi Cancer Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Masonic Cancer Center University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NEXT Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No